CLINICAL TRIAL: NCT01565980
Title: A Mindfulness Intervention for Symptom Management in Lung Cancer
Brief Title: Mindfulness Therapy for Individuals With Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Rebecca Lehto, PhD, RN, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CTSI grant
Record Dates: First submitted 2012-03-22; First posted 2012-03-29 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Lung Cancer
Keywords: Lung cancer; mindfulness therapy; active treatment (radiation and/or chemotherapy)
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- symptom assessment (Active Comparator): 6 weeks of symptom assessment phone calls.
  Interventions: Behavioral: symptom assessment
- Mindfulness intervention (Experimental): Participants receive 6 weeks of the home-based mindfulness intervention, and weekly symptom assessment phone calls.
  Interventions: Behavioral: symptom assessment; Behavioral: Mindfulness Intervention

INTERVENTIONS:
Behavioral: symptom assessment — attention control receives a weekly symptom assessment phone interview for 6 weeks.
Behavioral: Mindfulness Intervention — Participants will receive a weekly home-based mindfulness intervention, and symptom assessment phone interviews for 6 weeks.
  Arms: Mindfulness intervention

SUMMARY:
Managing psychological and physical symptoms to improve quality of life in patients with lung cancer are a major public health concern. Mindfulness-based therapies are showing promise in modifying psychological distress and improving quality of life in some cancer groups, but little testing has included lung cancer samples. Mindfulness-based therapies integrate meditation, breathing, and gentle yoga practices to promote an attitude of nonjudgmental acceptance and awareness of bodily states. Such strategies may promote well being, self-regulation, and symptom management. The study purpose was to test the acceptability, feasibility, and symptom / health-related quality of life (HRQOL) outcomes of a home-based mindfulness intervention for individuals with advanced lung cancer during non-curative treatment (radiation and/or chemotherapy). Acceptability and feasibility were measured via patient consent and retention rates, therapy expectancy, study adherence, attrition reasons, and quality assurance indicators. Efficacy was determined via symptom and HRQOL (health perceptions, physical and emotional function) outcomes. 40 patients undergoing treatment of non-small cell lung cancer were randomized to receive either six weekly mindfulness sessions (N=20) or an attention control condition (N=20). Outcome data was obtained at baseline (Time 1), post-intervention (Time 2, week 8), and four weeks after completion (Time 3, week 11). In addition, both groups received weekly symptom assessment interviews. The hypothesis was that the mindfulness group would report better symptom management and HRQOL (lower worry, dyspnea, insomnia, depression; higher physical and social function; more positive health perceptions) than the attention control group at the protocol end and that these differences will be sustained at Time 3.

DETAILED DESCRIPTION:
The final sample (n = 32) included 16 patients in the intervention and 16 in the attention control group (study attrition (n = 8, 20%).

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and speak English
2. at least 21 years old
3. active treatment for a diagnosis of non-small cell lung cancer
4. Karnofsky score > 80
5. have a telephone by which they can be reached

Exclusion Criteria:

1. current substance abuse other than tobacco
2. active treatment for psychiatric disorders excluding depression, and/or use of antipsychotic medications that would impede study participation.
3. cognitive impairment
4. active participation in mindfulness-based classes, guided imagery, yoga, or relaxation therapy courses
5. diagnosis of small cell lung cancer

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Lehto, PhD, Principal Investigator — Michigan State University
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Michigan State University, East Lansing, Michigan
  - Allegiance Health, Jackson, Michigan

REFERENCES:
- [Derived] Lehto RH, Wyatt G, Sikorskii A, Tesnjak I, Kaufman VH. Home-based mindfulness therapy for lung cancer symptom management: a randomized feasibility trial. Psychooncology. 2015 Sep;24(9):1208-12. doi: 10.1002/pon.3755. Epub 2015 Jan 28. No abstract available. PMID 25631362

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from two community-based hospital sites and one cancer center located in Chicago Illinois. Recruitment occurred between March 2012 to February 2013.
Pre-assignment Details: There were no participants excluded from the trial before group assignment. However, there were patients who dropped from the study before starting the intervention.
Groups:
- Symptom Assessment: weekly phone calls.
  symptom assessment: attention control group
- Mindfulness Intervention: Participants will receive 6 weeks of home-based mindfulness intervention.
  Mindfulness Intervention: Participants will receive a weekly home-based mindfulness intervention.
  Participants also receive weekly symptom assessment phone interview.
Period: Overall Study
Arm/Group | Symptom Assessment | Mindfulness Intervention
Started | 20 | 20 (Three patients had started the intervention protocol at the time of study withdrawal.)
Completed | 16 | 16
Not Completed | 4 | 4
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — health complications | 1 | 1
Not completed — stopped medical treatment | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Attention Control: weekly symptom assessment phone calls.
- Mindfulness Intervention: Participants receive weekly symptom assessment phone calls.
  Mindfulness Intervention: Participants receive 6 weekly sessions of a home delivered mindfulness intervention.
- Total: Total of all reporting groups
Arm/Group | Attention Control | Mindfulness Intervention | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (9.5) | 64.5 (9.25) | 66.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 17 | 19 | 36
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 16 | 18 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: M.D. Anderson Symptom Inventory (MDASI)
Description: Symptom Severity and interference were measured with the M.D. Anderson Symptom Inventory (MDASI) . The MDASI is a multisymptom patient-reported outcome measure. The MDASI has 13 core items include symptoms found to have the highest frequency and/or severity in patients with various cancers and treatment types (pain, fatigue, nausea, vomiting, disturbed sleep, distress, shortness of breath, memory difficulties, lack of appetite, drowsiness, dry mouth, sadness,numbness and tingling. Patients rate the severity of each symptom "at its worst" using 0-10 numerical rating scales with 0 = "not present" and 10 = "as bad as you can imagine." The measure includes 5 symptom interference items which ask how much all symptoms, interfere with domains (walking, work, general activity, mood, relations with others, enjoyment of life) also rated on a 0-10 scale (0 = "did not interfere"; 10 = "interfered completely"). The 13 severity (range 0 - 130) and 5 interference items (range 0 - 50) are summed.
Time Frame: Time 2 (week 8), Time 3 (week 11), and overall average for group comparisons.
Population: Adjusted means of outcomes and their standard errors are reported for times 2 and 3. The summary of linear mixed effects for group comparisons are then presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Attention Control Group: weekly phone calls.
  symptom assessment interview.
- Mindfulness Intervention: Participants receive 6 weekly sessions of a home delivered mindfulness intervention.
  Participants receive weekly phone calls to assess symptoms.
Arm/Group | Attention Control Group | Mindfulness Intervention
Number analyzed (Participants) | 16 | 16
units on a scale
  Symptom Severity - Time 2 | 33.91 (3.94) | 20.91 (4.30)
  Symptom Severity - Time 3 | 33.04 (3.98) | 22.86 (4.33)
  Symptom Severity - Summary | 32.11 (2.64) | 26.79 (2.84)
  Symptom Interference - Time 2 | 22.38 (2.63) | 10.45 (2.88)
  Symptom Interference - Time 3 | 19.27 (2.65) | 11.06 (2.90)
  Symptom Interference - Summary | 18.95 (1.74) | 4.33 (1.87)
Statistical Analysis 1: Comparison: Attention Control Group vs Mindfulness Intervention; The outcome measure was analyzed using linear mixed effects models (LME). The main effect of the trial arm was evaluated by averaging time 2 and time 3 values of the outcomes within the LME model. The resulting least square (LS) means and their standard errors are reported; Test type: Superiority or Other; p < .05, Mixed Models Analysis — P-values for the comparison of least square (LS) means represent the effect of the trial arm. The effect sizes are calculated as Cohen's d: difference between LS means divided by the standard deviation

2. Primary Outcome: SF-36
Description: Health-related Quality of Life (HRQOL) Indices (Physical/Emotional Function, Role Function, Pain, General Health, Vitality, Mental/Physical Health)HRQOL(SF-36) calculated using Quality Metric, Inc. an algorithm producing normal scores (1-100 range). With normed scoring, general population has mean=50, SD=10. For the minimum and maximum values in each of the scale ranges provided, higher values represent a better outcome.
Time Frame: Time 2 (week 8), Time 3 (week 11), and overall average for group comparisons.
Population: Adjusted means of outcomes and standards error provided for T2 & 3, folllowed by summary of linear mixed effects models for the outcomes for group comparisons.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Attention Control Group | Mindfulness Intervention
Number analyzed (Participants) | 16 | 16
units on a scale
  Physical Function -Time 2 | 34.94 (1.94) | 42.49 (2.02)
  Physical Function - Time 3 | 36.86 (1.94) | 43.31 (2.02)
  Physical Function - Summary | 35.90 (1.73) | 42.90 (1.82)
  Physical Role Function - Time 2 | 39.56 (2.22) | 41.61 (2.37)
  Physical Role Function - Time 3 | 41.82 (2.27) | 44.34 (2.37)
  Physical Role Function - Summary | 40.69 (1.80) | 42.97 (1.91)
  Bodily Pain Time 2 | 44.81 (2.52) | 51.22 (2.67)
  Bodily Pain Time 3 | 45.15 (2.56) | 46.58 (2.69)
  Bodily Pain Summary | 44.93 (2.25) | 48.89 (2.39)
  General Health - Time 2 | 46.05 (1.90) | 48.20 (2.04)
  General Health Summary | 44.59 (1.70) | 46.35 (1.82)
  Vitality Time 2 | 44.88 (2.19) | 47.49 (2.34)
  Vitality Time 3 | 43.37 (2.21) | 48.34 (2.34)
  Vitality Summary | 44.15 (2.06) | 47.92 (2.19)
  Social Function - Time 2 | 39.88 (2.22) | 47.54 (2.38)
  Social Function - Time 3 | 42.53 (2.28) | 48.97 (2.38)
  Social Function - Summary | 41.20 (1.75) | 48.25 (1.86)
  Emotional Role Function - Time 2 | 49.28 (1.78) | 51.15 (1.93)
  Emotional Role Function - Time 3 | 49.49 (1.82) | 51.40 (1.94)
  Emotional Role Function - Summary | 49.38 (1.68) | 51.28 (1.82)
  Mental Health - Time 2 | 49.61 (2.20) | 54.51 (2.35)
  Mental Health - Time 3 | 48.30 (2.22) | 54.51 (2.35)
  Mental Health - Summary | 48.97 (2.09) | 54.52 (2.23)
  Physical Overall - Time 2 | 37.14 (2.05) | 42.79 (2.16)
  Physical Overall - Time 3 | 38.29 (2.05) | 41.66 (2.16)
  Physical Overall - Summary | 37.72 (1.84) | 42.22 (1.96)
  Mental Overall - Time 2 | 50.72 (2.16) | 54.27 (2.29)
  Mental Overall - Time 3 | 49.84 (2.14) | 54.94 (2.29)
Statistical Analysis 1: Comparison: Attention Control Group vs Mindfulness Intervention; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — P values below 0.05 are considered statistically significant in this study

3. Other Pre Specified Outcome: Center for Epidemiologic Studies Depression (CES-D)
Description: The score is the sum of the 20 questions. Each item has a range of 1 - 4 for frequency of a behavior or mental state in the past week ; 1 - Rarely or none of the time (less than 1 day); 2 = Some or a little of the time (1-2 days); 3 = Occasionally or a moderate amount of time (3-4 days); 4 = Most or all of the time (5-7 days). Possible range is 0-60. There are 4 reverse-scored items (questions 4, 8, 12, and 16). A score of 16 points or more is considered depressed.
Time Frame: Time 2 (week 8), Time 3 (week 11), and overall average for group comparisons.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Attention Control Group | Mindfulness Intervention
Number analyzed (Participants) | 16 | 16
units on a scale
  CESD - Time 2 | 12.70 (1.84) | 8.07 (1.97)
  CESD - Time 3 | 12.83 (1.84) | 7.63 (1.97)
  CESD - Summary | 12.76 (1.68) | 7.84 (1.80)
Statistical Analysis 1: Comparison: Attention Control Group vs Mindfulness Intervention; Test type: Superiority or Other; p < .05, Mixed Models Analysis — P values below 0.05 are considered statistically significant in this study

4. Other Pre Specified Outcome: Cancer Dyspnea Scale
Description: The cancer dyspnea scale (CDS) has 12 Likert scale items ( 1 = Not at all, 5 = Very much) that ask questions about breathlessness or difficulty in breathing during the past few days. The CDS has an overall score (range 0-42) and 3 subscales that measure the amount of effort with breathing, anxiety associated with breathing, and discomfort associated with breathing.
  The 3 subscales are calculated by: 1) effort (items 4+6+8+10+12) - 5 [range 0 (no dyspnea effort)-20 (worst dyspnea effort)]; 2) anxiety (items 5+7+9+11) - 4 [range 0 (no dyspnea anxiety) - 16 (worst dyspnea anxiety)]; 3) discomfort [15 - (items 1+2+3) {range 0 (no dyspnea discomfort) - 12 (worst dyspnea discomfort)}]. The total dyspnea score is derived by adding the total subscale scores. The subscale score subtractions are to make adjustments for 0 as a state of absence of dyspnea (thus total dyspnea summary scores range from 0 to 42).
Time Frame: Time 2 (week 8), Time 3 (week 11), and overall average for group comparisons.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Attention Control Group | Mindfulness Intervention
Number analyzed (Participants) | 16 | 16
units on a scale
  CDS total score - Time 2 | 7.69 (1.10) | 4.07 (1.19)
  CDS total score - Time 3 | 7.50 (1.10) | 3.21 (1.19)
  CDS - total score - Summary | 7.60 (.99) | 3.64 (1.07)
  CDS - effort - Time 2 | 4.25 (.54) | 2.06 (.58)
  CDS - effort - Time 3 | 4.44 (.54) | 2.14 (.59)
  CDS - effort - summary | 4.34 (.50) | 2.10 (.54)
  CDS - anxiety - Time 2 | .93 (.40) | .79 (.43)
  CDS - anxiety - Time 3 | .80 (.40) | .58 (.43)
  CDS - anxiety - summary | .87 (.32) | .69 (.34)
  CDS - discomfort - Time 2 | 2.80 (.56) | .87 (.60)
  CDS - discomfort - Time 3 | 2.55 (.56) | .16 (.60)
  CDS - discomfort - summary | 2.68 (.48) | .51 (.52)
Statistical Analysis 1: Comparison: Attention Control Group vs Mindfulness Intervention; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — P values below 0.05 are considered statistically significant in this study

5. Other Pre Specified Outcome: Worry (Cancer-related and General)
Description: Both cancer-related and general worry were measured with 3 item scales. Cancer-related worry had three statements asking about level of worry related to diagnosis, treatment, and worry interference using a 1 = "not at all" to 5 = "most or all the time" scale, range 3-15. Items are summed. General worry used an abbreviated brief Penn State Worry questionnaire with 3 statements that measure how typical that statements are in describing the person. Uses a 3 item scale with 1 = "not at all typical" to 5 = "very typical". the range is 3-15. Items are summed.
Time Frame: Time 2 (week 8), Time 3 (week 11), and overall average for group comparisons.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Attention Control Group | Mindfulness Intervention
Number analyzed (Participants) | 16 | 16
units on a scale
  Cancer-related worry - Time 2 | 8.26 (.58) | 6.28 (.62)
  Cancer-related worry - Time 3 | 7.88 (.58) | 6.06 (.62)
  Cancer-related worry - Summary | 8.07 (.49) | 6.17 (.53)
  General worry - Time 2 | 5.89 (.52) | 5.41 (.56)
  General worry - Time 3 | 7.88 (.58) | 6.06 (.62)
  General worry - Summary | 8.07 (.49) | 6.17 (.53)
Statistical Analysis 1: Comparison: Attention Control Group vs Mindfulness Intervention; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — P values below 0.05 are considered statistically significant in this study

6. Other Pre Specified Outcome: Pittsburgh Sleep Symptom Questionnaire-Insomnia (PSSQ_I)
Description: The PSSQ_I has 13 self rated questions. The first 5 items, used to determine sleep quality (presence; frequency of insomnia problems) are rated [0 = never to 5 = always, 5-7 days per week; (range 0-25)] and items 6 to 13 are aimed at identifying the degree of interference experienced from sleep impairment (rated 0=not at all to 4=extremely on Likert scale; range 0 - 32).
Time Frame: Time 2 (week 8), Time 3 (week 11), and overall average for group comparisons.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Symptom Assessment | Mindfulness Intervention
Number analyzed (Participants) | 16 | 16
units on a scale
  PSSQ_I Quality -Time 2 | 10.62 (1.95) | 8.71 (2.14)
  PSSQ_I Quality-Time 3 | 12.93 (1.99) | 8.17 (2.08)
  PSSQ_I Quality- Overall | 11.76 (1.75) | 8.38 (1.87)
  PSSQ_I Interference- Time 2 | 6.45 (1.47) | 5.99 (1.55)
  PSSQ_I Interference- Time 3 | 9.26 (1.54) | 6.28 (1.55)
  PSSQ_I Interference- Overall | 7.80 (1.25) | 6.13 (1.29)
Statistical Analysis 1: Comparison: Symptom Assessment vs Mindfulness Intervention; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — P values below 0.05 are considered statistically significant in this study

7. Other Pre Specified Outcome: Baseline Values for All Measures.
Description: Description of all measures are described elsewhere. Provided are the means and standard deviations for baseline comparisons.
Time Frame: Baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Symptom Assessment | Mindfulness Intervention
Number analyzed (Participants) | 16 | 16
units on a scale
  MDASI Symptom Severity (range 0-130) | 29.25 (19.18) | 35 (21.26)
  MDASI Symptom Interference (range 0-50) | 19.15 (16.41) | 21.25 (16.2)
  HRQOL -Physical Function (range 0-100) | 35.25 (10.17) | 37.73 (8.90)
  HRQOL - Physical Role Function (range 0-100) | 40.31 (10.47) | 38.97 (9.64)
  HRQOL - Bodily Pain (range 0-100) | 47.36 (12.29) | 41.96 (9.59)
  HRQOL - General Health (range 0-100) | 46.43 (11.66) | 41.89 (11.60)
  HRQOL - Vitality (range 0-100) | 45.91 (11.96) | 42.2 (7.5)
  HRQOL - Social Function (range 0-100) | 47.56 (10.72) | 41.55 (11.42)
  HRQOL - Emotional Function(range 0-100) | 47.12 (12.75) | 46.77 (11.25)
  HRQOL - Mental Health (range 0-100) | 49.56 (10.13) | 45.37 (10.07)
  HRQOL - Physical Summary (range 0-100) | 39.17 (10.43) | 37.83 (8.91)
  HRQOL - Mental Summary (range 0-100) | 51.82 (12.23) | 47.33 (11.01)
  CESD - Depression (range 0-60) | 10.35 (8.27) | 15.9 (10.51)
  CDS - Overall Dyspnea (range 0-42) | 8.85 (8.86) | 7.05 (6.23)
  CDS - Effort (range 0-20) | 4.85 (4.98) | 4.45 (4.47)
  CDS - Anxiety (range 0-16) | 1.55 (2.72) | .85 (1.5)
  CDS - Discomfort (range 0-12) | 2.45 (2.63) | 1.75 (1.97)
  Worry - General (range 3-15) | 5.55 (3.09) | 7.35 (4.07)
  Worry - Cancer-related (range 3-15) | 7.45 (3.63) | 9.70 (3.57)
  PSSQ_I Sleep quality (range 0-25) | 11.65 (7.53) | 14.47 (6.84)
  PSSQ_I Sleep interference (range 0-32) | 6.37 (6.18) | 10.63 (8.05)
Statistical Analysis 1: Comparison: Symptom Assessment vs Mindfulness Intervention; Test type: Superiority or Other; p < 0.05, Descriptive statistics for outcomes — P values above 0.05 are considered statistically insignificant in this study

ADVERSE EVENTS:
Time Frame: 1 year.
Groups:
- Mindfulness Intervention: Participants will receive 6 weeks of home-based mindfulness intervention.
  Mindfulness Intervention: Participants will receive a weekly home-based mindfulness intervention.
Arm/Group | Symptom Assessment | Mindfulness Intervention
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No